CLINICAL TRIAL: NCT02235116
Title: Predictors of Patient Attitudes and Barriers to Skin Cancer Screening
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-001705
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2014-09

CONDITIONS: Skin Cancer
Keywords: Number of patients; full body skin exam; Survey; preferences
MeSH Terms: conditions — Skin Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who responded to the survey
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
This is a cross-sectional survey distributed to a convenience sample of patients in a waiting room of an academic dermatology clinic. The survey assesses patient experiences with full body skin exams and attitudes towards full body skin exams. The survey is designed to help investigators better understand how many patients are not getting full body skin exams, why this may be occurring, and what types of interventions may be enacted to increase the number of patients getting full body skin exams.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* English-speaking

Exclusion Criteria:

* previously completed the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: English-speaking patients 18yrs old and older attending the UCLA Dermatology clinics in Santa Monica, California or Westwood, California from June 14 to July 1, 2011
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of patients reporting ever having had a full body skin examination | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Chiu, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Dermatology, Los Angeles, California, United States